CLINICAL TRIAL: NCT04323657
Title: Phase 1/2 Trial of TC-110 T Cells in Adults With Relapsed or Refractory Non-Hodgkin Lymphoma (NHL) or Acute Lymphoblastic Leukemia (ALL)
Brief Title: TC-110 T Cells in Adults With Relapsed or Refractory Non-Hodgkin Lymphoma or Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TCR2 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCR2-19-01
Record Dates: First submitted 2020-03-22; First posted 2020-03-26 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Non Hodgkin Lymphoma; Acute Lymphoblastic Leukemia; Diffuse Large B Cell Lymphoma; Primary Mediastinal Large B Cell Lymphoma; Mantle Cell Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): The Phase 1 portion of the study will proceed according to a standard 3 + 3 dose escalation schema. Patients will be enrolled into 3 cohorts based on disease: NHL cohort, low tumor burden ALL cohort, and high tumor burden ALL cohort.
  Interventions: Drug: TC-110 T Cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 2 (Experimental): The phase 2 portion of the study will evaluate the efficacy of TC-110 T cells administered at the RP2D, preceded by a lymphodepleting regimen.
  Interventions: Drug: TC-110 T Cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: TC-110 T Cells — TC-110 T Cells
Drug: Fludarabine — Flu/Cy Lymphodepletion
Drug: Cyclophosphamide — Flu/Cy Lymphodepletion

SUMMARY:
TC-110 T cells are a novel cell therapy that consists of autologous genetically engineered T cells expressing a single-domain antibody that recognizes human CD19, fused to the CD3-epsilon subunit which, upon expression, is incorporated into the endogenous T cell receptor (TCR) complex.

This is a Phase 1/2 open-label study to evaluate the safety of autologous genetically engineered TC-110 T cells in patients with aggressive NHL (DLBCL, PMBCL, TFL), high-risk indolent NHL (including MCL), or adult ALL.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years of age at the time the Informed Consent is signed
* Patient has agreed to abide by all protocol-required procedures, including study-related assessments, and management by the treating institution for the duration of the study and LTFU
* Histologically confirmed NHL or ALL
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Patient must have adequate organ function as indicated by the laboratory values in the clinical protocol
* Patient must be fit for leukapheresis and have adequate venous access for cell collection
* Patient must have evidence of CD19 expression
* Prior CD19-directed CAR T therapy is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Establish the recommended phase 2 dose (RP2D) for the NHL and ALL indications according to the observed adverse events, including potential dose-limiting toxicities (DLT). | DLTs within 28 days post-treatment
To evaluate the efficacy of autologous genetically modified TC-110 T cells in adult patients with R/R NHL as determined by overall response rate (ORR) | ORR at 3 months for NHL patients at 3 months
To evaluate the efficacy of autologous genetically modified TC-110 T cells in adult patients with R/R ALL as determined by overall response rate and Minimum Residual Disease (MRD) negativity rates | ORR rate and MRD negativity rate for ALL patients at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical, Study Chair — TCR2 Therapeutics
Locations (3):
- United States (3):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No